CLINICAL TRIAL: NCT05136625
Title: Sphenopalatine Ganglion Block and Pain Management in Neurosurgery
Acronym: SpheNoPain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 553/2021/Sper/AOUFe
Record Dates: First submitted 2021-10-18; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-09

CONDITIONS: Post Operative Pain; Craniofacial Pain
Keywords: sphenopalatine ganglion block; post-craniotomy pain
MeSH Terms: conditions — Pain, Postoperative; Facial Pain | interventions — Sphenopalatine Ganglion Block; Reference Standards

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Troncular scalp blockade (Levobupivacaine 7,5%) Local site infiltration (Mepivacaine)
  Interventions: Drug: Standard Preparation
- Treatment (Experimental): Troncular scalp blockade (Levobupivacaine 7,5%) Local site infiltration (Mepivacaine) Transnasal sphenopalatine ganglion block (Levobupivacaine 7,5%)
  Interventions: Drug: Sphenopalatine ganglion block; Drug: Standard Preparation

INTERVENTIONS:
Drug: Sphenopalatine ganglion block — A cotton swab soaked in levobupivacaine 7,5% in inserted into the nose to block sphenopalatine ganglion, with the classic technique previously described
  Arms: Treatment
Drug: Standard Preparation — Troncular scalp blockade. Local site infiltration

SUMMARY:
Post craniotomy pain is defined as headache developed up to 7 days from a craniotomy, not otherwise explained. A moderate to severe pain affects from 60 to 84% of patients.

Sphenopalatine ganglion block has been successfully used in patients with chronic or acute headache, facial pain and for transsphenoidal pituitary and endoscopic sinus surgeries.

There are evidences that sphenopalatine ganglion block reduces vegetative responses to skull pin closure.

This study aim to investigate feasibility and efficacy of sphenopalatine ganglion block in reducing pain after a neurosurgical supratentorial craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* supratentorial craniotomy

Exclusion Criteria:

* prior craniofacial pain syndrome
* drug assumption: pain-killers (chronic), antiepileptic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Immediately post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 1° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 2° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 3° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 4° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 30° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 60° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Numerical Rating Scale | 180° days post-op
  From 0 (no pain) to 10 (worst pain ever)
Visual Analogic Scale | Immediately post-op
  From 0 (no pain) to 10 (worst pain ever)
Visual Analogic Scale | 1° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 2° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 3° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 4° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 30° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 60° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Visual Analogic Scale | 180° day post-op
  From 0 (no pain) to 10 (worst pain ever) on a straight line
Pain Assessment IN Advanced Dementia | Immediately post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 1° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 2° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 3° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 4° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 30° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 60° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)
Pain Assessment IN Advanced Dementia | 180° day post-op
  From 0 (no signs of pain) to 10 (Extreme pain)

SECONDARY OUTCOMES:
Adverse effect | Immediately post-op, 1°-2°-3°-4°-30°-60°180° days post-op
  Bitter taste, nose bleeding, throat discomfort
Vegetative response (Heart rate) | 1-5-10 min from skull pin closure. 1-5-10 min from skin incision
  Heart rate in beat per minute
Vegetative response (Arterial pressure) | 1-5-10 min from skull pin closure. 1-5-10 min from skin incision
  Mean arterial pressure in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale De Bonis, MD PhD, Study Chair — Università degli Studi di Ferrara
Locations (1):
- Sant'Anna Hospital, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sir E, Eksert S. Morphological Description and Clinical Implication of Sphenopalatine Foramen for Accurate Transnasal Sphenopalatine Ganglion Block: An Anatomical Study. Medeni Med J. 2019;34(3):239-243. doi: 10.5222/MMJ.2019.20586. Epub 2019 Sep 27. PMID 32821444
- [Background] Padhy N, Moningi S, Kulkarni DK, Alugolu R, Inturi S, Ramachandran G. Sphenopalatine ganglion block: Intranasal transmucosal approach for anterior scalp blockade - A prospective randomized comparative study. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):207-212. doi: 10.4103/joacp.JOACP_249_18. Epub 2020 Jun 15. PMID 33013036
- [Background] Crespi J, Bratbak D, Dodick D, Matharu M, Jamtoy KA, Aschehoug I, Tronvik E. Measurement and implications of the distance between the sphenopalatine ganglion and nasal mucosa: a neuroimaging study. J Headache Pain. 2018 Feb 13;19(1):14. doi: 10.1186/s10194-018-0843-5. PMID 29442191
- [Background] Elahi F, Ho KW. Successful Management of Refractory Headache and Facial Pain due to Cavernous Sinus Meningioma with Sphenopalatine Ganglion Radiofrequency. Case Rep Neurol Med. 2014;2014:923516. doi: 10.1155/2014/923516. Epub 2014 Sep 29. PMID 25343051
- [Derived] Mantovani G, Sgarbanti L, Indaimo A, Cavallo MA, De Bonis P, Flacco ME, Scerrati A. Effects of a sphenopalatine ganglion block on postcraniotomy pain management: a randomized, double-blind, clinical trial. Neurosurg Focus. 2023 Dec;55(6):E13. doi: 10.3171/2023.9.FOCUS23549. PMID 38262005